CLINICAL TRIAL: NCT02131714
Title: Pressure Pain Threshold of Jaw Muscles in Patients With Facial Myofascial Pain Submitted to a Conservative Treatment : a Short-term Evaluation
Brief Title: Pressure Pain Threshold of Jaw Muscles in TMD Patients Submitted to a Conservative Treatment
Acronym: PPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Monique Lalue Sanches, DDS, Federal University of São Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMD-2003
Record Dates: First submitted 2014-04-21; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Pain; Myofascial Pain; Temporomandibular Disorder Syndrome; Therapeutic Exercise; Facial Pain
Keywords: pressure pain threshold; temporomandibular disorder syndrome; therapeutic exercise; conservative treatment; facial pain
MeSH Terms: conditions — Pain; Facial Pain | interventions — Counseling; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- counseling and exercises (Active Comparator): These individuals were asked about parafunctional habits and the treatment was applied by providing an explanation concerning the role of pain, possible aetiological factors of the patient's TMD, the relationship between chronic pain and psychosocial distress, and its benign character. They also had to perform once daily application of hot packs on both sides of the face for 20 minutes and after that they must perform active free therapeutic exercise of mouth opening for 10 times
  Interventions: Behavioral: counseling and exercises
- lifestyle counseling (Placebo Comparator): These individuals were asked about parafunctional habits and the treatment was applied by providing an explanation concerning the role of pain, possible aetiological factors of the patient's TMD, the relationship between chronic pain and psychosocial distress, and its benign character.
  Interventions: Behavioral: lifestyle counseling

INTERVENTIONS:
Behavioral: counseling and exercises — These individuals were asked about parafunctional habits and the treatment was applied by providing an explanation concerning the role of pain, possible aetiological factors of the patient's TMD, the relationship between chronic pain and psychosocial distress, and its benign character. They also had to perform once daily application of hot packs on both sides of the face for 20 minutes and after that they must perform active free therapeutic exercise of mouth opening for 10 times
  Arms: counseling and exercises
Behavioral: lifestyle counseling
  Arms: lifestyle counseling

SUMMARY:
Pain is an unpleasant sensory and emotional experience that is one of the main symptoms of temporomandibular disorder (TMD). One way to assess pain is through algometry. The aim of this study was to evaluate, by the pressure pain threshold measurements, the efficacy of a short-term conservative treatment for the management of temporomandibular disorders. This study is a randomized controlled clinical trial where 84 participants were diagnosed with myofascial pain according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD), with a mean age of 44 years old ranging from 18 to 76 years old. These individuals were asked about parafunctional habits and the treatment was applied by providing an explanation concerning the role of pain, possible aetiological factors of the patient's TMD, the relationship between chronic pain and psychosocial distress, and its benign character. They also had to perform once daily application of hot packs on both sides of the face for 20 minutes and after that they must perform active free therapeutic exercise of mouth opening for 10 times. The pressure pain threshold of the masseter and temporalis muscles and the lateral pole of the condyle were obtained at baseline (T0), between 15 and 30 days after (T1) and at 75 to 90 days after (T2) representing the end of the treatment. Two groups of subjects were obtained. The first was considered the study group (SG) and included those who underwent the treatment proposed. The control group (CG) consisted of participants who did not undergo treatment because they did not believe in it.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old have diagnosis of myofascial pain according RDC/TMD signed the informed consent

Exclusion Criteria:

* people under 18 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
pressure pain threshold (PPT) in Kilogram-force (Kgf) | at baseline (first appointment)
  -pressure pain threshold (PPT) from masseter and temporalis muscles, and lateral pole of the condyle in both sides of the face.
  It was measured with a digital algometer.
pressure pain threshold (PPT) in Kilogram-force (Kgf) | 3 to 4 weeks (second appointment)
  -pressure pain threshold (PPT) from masseter and temporalis muscles, and lateral pole of the condyle in both sides of the face.
  It was measured with a digital algometer.
pressure pain threshold (PPT) in Kilogram-force (Kgf) | 10 to 12 weeks (last appointment)
  pressure pain threshold (PPT) from masseter and temporalis muscles, and lateral pole of the condyle in both sides of the face.
  It was measured with a digital algometer.

SECONDARY OUTCOMES:
Visual analogue scale (VAS). A line with 100mm where in one extremity its wrote "no pain" and in the end of the line its wrote "the worst pain" | at baseline (first appointment)
  - Visual analogue scale (VAS) for measuring pain.
Verbal numerical scale (VNS) is a 11- point scale (0 to 10) | at baseline (first appointment)
  - Verbal numerical scale (VNS) for measuring pain. Ask the patient to quantify his pain in a 11-point pain scale, where 0 is no pain and 10 the worst pain he ever had.
Visual analogue scale (VAS). A line with 100mm where in one extremity its wrote "no pain" and in the end of the line its wrote "the worst pain" | 3 to 4 weeks (second appointment)
  Visual analogue scale (VAS) for measuring pain.
Visual analogue scale (VAS). A line with 100mm where in one extremity its wrote "no pain" and in the end of the line its wrote "the worst pain" | 10 to 12 weeks (last appointment)
  Visual analogue scale (VAS) for measuring pain.
Verbal numerical scale (VNS) is a 11- point scale (0 to 10) | 3 to 4 weeks (second appointment)
  Verbal numerical scale (VNS) for measuring pain. Ask the patient to quantify his pain in a 11-point pain scale, where 0 is no pain and 10 the worst pain he ever had.
Verbal numerical scale (VNS) is a 11- point scale (0 to 10) | 10 to 12 weeks (last appointment)
  Verbal numerical scale (VNS) for measuring pain. Ask the patient to quantify his pain in a 11-point pain scale, where 0 is no pain and 10 the worst pain he ever had.

OTHER OUTCOMES:
oral health impact profile - (OHIP-14) modified | at baseline (first appointment)
  It's a questionnaire to avaliate the impact profile of his temporomandibular joint condition and pain on his lifestyle.
Catastrophizing scale of the coping strategies questionnaire (CSQ) | at baseline (first appointment)
  CSQ - coping strategies questionnaire To avaliate how catastrophizing toughts are present before and after treatment protocol was applied.
oral health impact profile - (OHIP-14) modified | 10 to 12 weeks (last appointment)
  It's a questionnaire to avaliate the impact profile of his temporomandibular joint condition and pain on his lifestyle.
Catastrophizing scale of the coping strategies questionnaire (CSQ) | 10 to 12 weeks (last appointment)
  CSQ - coping strategies questionnaire To avaliate how catastrophizing toughts are present before and after treatment protocol was applied.

CONTACTS AND LOCATIONS:
Overall Officials: Luis G Alonso, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Ambulatorio de Disfunção Temporomandibular e Dor Orofacial, São Paulo, São Paulo, Brazil